CLINICAL TRIAL: NCT07053514
Title: Same-Day Antiretroviral Therapy as a Behavioral Design Intervention to Reduce Stigma in Key Affected Populations
Acronym: Peru SD-ART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000040491; R01TW013180 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: PWH in Peru and HIV clinicians prescribing ART.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People With HIV (PWH) (Experimental): SD-ART protocol for PWH prescribed by their HIV clinicians
  Interventions: Behavioral: SD-ART
- Clinicians prescribing ART (No Intervention)

INTERVENTIONS:
Behavioral: SD-ART — SD-ART protocol for PWH with both patients and their HIV clinicians
  Arms: People With HIV (PWH)

SUMMARY:
The goal of this study is to develop and implement a same-day ART (SD-ART) protocol for key affected populations with HIV in Peru. The development of the protocol will be guided by asynchronous online focus groups with HIV experts to define eligibility criteria and essential components of the protocol, as well as nominal group technique focus groups and in-depth interviews to identify barriers and facilitators to SD-ART implementation. Finally, investigators will pilot the SD-ART protocol with patients and clinicians using a prospective, longitudinal design integrated into routine HIV care.

DETAILED DESCRIPTION:
The proposed study has 3 aims:

1. Conduct asynchronous online focus groups (AOFGs) and flowcharting to map the current ART initiation process and design a streamlined same-day antiretroviral therapy (SD-ART) protocol as a behavioral design.
2. Assess the multi-level barriers and facilitators to refine and implement an SD-ART protocol from the perspectives of patients, clinicians, and administrators, considering the high levels of stigma and suboptimal HIV treatment outcomes. Findings from Aims 1 and 2 will guide Aim 3.
3. Pilot-test the protocol-concordant SD-ART strategy in newly diagnosed People with HIV where investigators will assess and follow multi-level stigma constructs in patients and providers, analyzed through longitudinal dyadic analyses, to provide the evidence for SD-ART as a behavioral design intervention that reduces stigma.

The focus of this registration is the trial in aim 3.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1:

HIV experts will be selected from National Societies of HIV experts according to the following criteria: 1) 18 years old or older; 2) Be an HIV expert, including those from NGOs providing HIV care, and international specialists; 3) Provide informed consent.

* Aim 2:

  * NGT Focus Groups (FG)

    * Staff members

      1. 18 years old or older.
      2. Be a clinical staff member at Hospital Dos de Mayo or Patrucco Primary Health Center.
      3. Provide informed consent.
    * PWH receiving HIV care

      1. 18 years old or older.
      2. Identify as member of a KAP.
      3. Receive HIV care at Hospital Dos de Mayo or Patrucco Primary Health.
      4. Provide informed consent.
    * PWH who dropped out of HIV care

      1. 18 years old or older.
      2. Identify as a member of a KAP.
      3. Previously received HIV care at Hospital Dos de Mayo or Patrucco Primary Health but dropped out of care, as identified through patient registries.
      4. Provide informed consent.
  * In-depth interviews

    * 1) 18 years old or older.
    * 2) Be the director of Hospital Dos de Mayo or Patrucco primary health center or the HIV director at the Ministry of Health
    * 3) Provide informed consent
* Aim 3:

  * Clinical Staff Dyadic Surveys

    * 1) 18 years old or older.
    * 2) Be an HIV provider at Hospital Dos de Mayo or Raul Patrucco Primary Health Center.
    * 3) Provide HIV care to one of the 125 PWH
    * 4) Provide informed consent.
  * Patient Dyadic Surveys

    * 1) 18 years old or older.
    * 2) Identify as a member of a KAP.
    * 3) Be newly diagnosed with HIV and eligible for SD-ART based on clinical criteria identified from Aims 1 and 2.
    * 4) Provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2027-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Reductions in patient HIV and multi-dimensional stigma | baseline, month 1, month 3, month 6, month 9, and month 12
  Assessed using a modified 10-item version of the Berger HIV stigma scale, which has been previously translated into Spanish and validated in Peru. Total score range from 40 to 160. Higher scores denote higher levels of HIV stigma.
Provider stigma toward patients | baseline, month 1, month 3, month 6, month 9, and month 12
  Measured through feeling thermometers (on a scale from 0-100) of various identity groups (people with HIV, sexual minorities, people who use drugs).
Everyday Discrimination Scale | baseline, month 1, month 3, month 6, month 9, and month 12
  This is a 5-item scale that is rated on a 6-point scale (range from 0 to 30), with higher scores denoting higher levels of multi-dimensional stigma and experiences with discrimination

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, M.D., M.A, Principal Investigator — Yale University
Locations (2):
- Peru (2):
  - Centro de Salud Raul Patrucco Puig, Lima
  - Hospital Dos de Mayo, Lima

IPD SHARING:
Plan to Share IPD: No